CLINICAL TRIAL: NCT05915494
Title: Intermittent Pneumatic Compression in Inhalation Injury: Effects on Diaphragm Mobility and Pulmonary Function in Children Sufferers
Brief Title: Intermittent-pneumatic Compression in Inhalation-injury Children: Effects on Diaphragm Mobility and Pulmonary Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Internal Medicine and Geriatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004529
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Inhalation Injury
MeSH Terms: interventions — Physical Therapy Modalities; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): intermittent pneumatic compression group (n = 20 inhalation injury children). in this children group, intermittent pneumatic compression will be used to resist diaphragm muscle during 10-set-training session which will be done five session per the week, for 12 weeks. besides this training, traditional physical therapy program will be handled). In other inhalation group, n =20, traditional physical therapy program will be handled only). Also, free walking for 30 minutes daily will be performed by children.
  Interventions: Other: intermittent pneumatic compression, physiotherapy, and walking
- group B (Active Comparator): traditional physiotherapy group (n = 20 inhalation injury children). In this inhalation group, traditional physical therapy program will be handled only for 12 weeks. Also, free walking for 30 minutes daily will be performed by children.
  Interventions: Other: physiotherapy and walking

INTERVENTIONS:
Other: intermittent pneumatic compression, physiotherapy, and walking — intermittent pneumatic compression group (n = 20 inhalation injury children). in this children group, intermittent pneumatic compression will be used to resist diaphragm muscle during 10-set-training session which will be done five session per the week, for 12 weeks. besides this training, traditional physical therapy program will be handled). In other inhalation group, n =20, traditional physical therapy program will be handled only). Also, free walking for 30 minutes daily will be performed by children.
  Arms: group A
Other: physiotherapy and walking — in this children group, n = 20, for 12 weeks, traditional physical therapy program (chest physical therapy, flexibility exercises, range of motion exercises) will be handled. Also, free walking for 30 minutes daily will be performed by children.
  Arms: group B

SUMMARY:
inhalation injury is very common in infants, young, children. complications of this problems are low pulmonary functions and limited mobility of main inspiratory muscle.

DETAILED DESCRIPTION:
inhalation injury patients (children, n = 40) will be included in intermittent pneumatic compression group (n = 20, this device, intermittent pneumatic compression, will be used a resistive inspiratory muscle training for diaphragm muscle and the 10-set training will be done five session per the week, for 12 weeks. besides this training, traditional physical therapy program will be handled). In other inhalation group, n =20, traditional physical therapy program will be handled only)

ELIGIBILITY:
Inclusion Criteria:

* inhalation injury

Exclusion Criteria:

* brain injury
* fractures of any body part
* cardiac or chest disorders

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — based on self-representation of birth-certificate identity.
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
forced vital capacity | it will be measured after 12 weeks
  it is a pulmonary function test

SECONDARY OUTCOMES:
forced expiatory volume at the first second of expiration | it will be measured after 12 weeks
  it is a pulmonary function test
right-side diaphragmatic excursion | it will be measured after 12 weeks
  it will be assessed by ultrasonographic measurements
left-side diaphragmatic excursion | it will be measured after 12 weeks
  it will be assessed by ultrasonographic measurements
upper chest expansion | it will be measured after12 weeks
  it will be assessed by tape
lower chest expansion | it will be measured after 12 weeks
  it will be assessed by tape

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt